CLINICAL TRIAL: NCT06039163
Title: A Randomized, Double-blind, Placebo-controlled, Phase 1 Study to Assess the Safety, Tolerability, Preliminary Efficacy of Inhaled HH-120 Aerosol in Participants With Mild to Moderate COVID-19
Brief Title: A Study to Assess the Safety, Tolerability and Preliminary Efficacy of HH-120 for the Treatment of COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Huahui Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HH120-103
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HH-120 (Active Comparator)
  Interventions: Drug: HH-120
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: HH-120 — Participants randomized to active treatment in escalation phase will receive HH-120 administered via inhalation for 5 consecutive days (Day 1 to Day 5). Planned dose levels to be used for the escalation phase of the study are 50 (BID), 50 (TID), and 100 (BID) mg. The expansion phase will begin once the recommended dose for expansion phase determined, based on safety and preliminary efficacy data from the escalation phase.
  Arms: HH-120
Drug: placebo — Participants randomized to placebo group in escalation and expansion phase will receive placebo administered via inhalation for 5 consecutive days (Day 1 to Day 5).
  Arms: placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled Phase 1 study in participants over the age of 18 years with mild to moderate COVID-19. This study aims to assess the safety, tolerability and preliminary antiviral effect of HH-120. This study includes dose escalation phase and dose expansion phase.

ELIGIBILITY:
Inclusion Criteria:

* The escalation phase:

  1. Participants are aged 18 to 65 years (inclusive at the time of informed consent)
  2. Participants are mild or moderate COVID-19 patients.
  3. Participants have one or more mild or moderate COVID 19-related symptoms as defined by the FDA (see the Diagnosis and Main Criteria for Inclusion) with the onset of symptoms ≤ 3 days prior to the randomization.
* The expansion phase:

  1. Participants are ≥18 years of age at the time of randomization.
  2. Participants are mild or moderate COVID-19 patients.
  3. Participants have one or more mild or moderate COVID 19-related symptoms as defined by the FDA (see the Diagnosis and Main Criteria for Inclusion) with the onset of symptoms ≤ 5 days prior to the randomization.

Exclusion Criteria:

* Pregnant or lactating at Screening or planning to become pregnant (self or partner) at any time during the study, including the follow-up period.
* Prior or ongoing medical conditions, medical history, physical findings, or laboratory abnormality that, in the PI's (or delegate's) opinion, could adversely affect the safety of the participant or that might interfere with the conduct of the study.
* Presence of any underlying physical or psychological medical condition that, in the opinion of the PI, would make it unlikely that the participant will comply with the protocol or complete the study per protocol.
* Have known allergies to any of the components used in the formulation of the study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-04-16 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability: Incidence, frequency, severity, and duration of treatment-emergent adverse events (TEAEs), treatment-related adverse events (TRAE) and serious adverse events (SAEs), etc. | From Baseline to Day 12

SECONDARY OUTCOMES:
Proportion of participants that achieve SARS-CoV-2 clearance (defined as negative qRT-PCR tests taken on two consecutive days), with the time of clearance being the time of the first negative test. | From Baseline to Day 12
Median time to achieve SARS-CoV-2 clearance (defined as negative qRT-PCR tests taken on two consecutive days), with the time of clearance being the time of the first negative test. | From Baseline to Day 12
Median time to sustained clinical recovery. | From Baseline to Day 12

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Beijing Ditan Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Guangzhou Eighth People's,Guangzhou Medical University, Guangzhou, Guangdong
  - The First Hospital of Jilin University, Changchun, Jilin
  - Huashan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality